CLINICAL TRIAL: NCT03062917
Title: Validation of Nasal and Bronchial Absorption Sampling Methods for the Assessment of RSV Bronchiolitis in Babies and Children
Brief Title: Nasal and Bronchial Absorption Sampling in RSV Bronchiolitis
Acronym: RSV-SAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College Healthcare NHS Trust (Other)
Collaborators: Pulmocide Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 15/WM/0343
Record Dates: First submitted 2017-02-07; First posted 2017-02-24 (Actual); Results first posted 2019-11-12 (Actual); Last update posted 2019-11-12 (Actual); Status verified 2019-10

CONDITIONS: Bronchiolitis; Bronchiolitis, Viral; RSV Infection; Respiratory Failure
MeSH Terms: conditions — Bronchiolitis; Bronchiolitis, Viral; Respiratory Syncytial Virus Infections; Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Emergency Department (Other): Babies with suspected respiratory tract infection (RTI) in the ED
  Interventions: Diagnostic Test: Nasal and Bronchial Sampling
- Paediatric Wards (Other): Babies with diagnosed RSV infection admitted to paediatric wards
  Interventions: Diagnostic Test: Nasal and Bronchial Sampling
- Paediatric Intensive Care (Other): Babies with diagnosed severe RSV infection in PICU requiring mechanical ventilation
  Interventions: Diagnostic Test: Nasal and Bronchial Sampling
- Health Controls (Other): Babies without respiratory symptoms, attending routine outpatient appointments or undergoing elective surgical procedures
  Interventions: Diagnostic Test: Nasal and Bronchial Sampling
- Controls in Paediatric Intensive Care (Other): Babies without RSV infection but requiring mechanical ventilation in PICU
  Interventions: Diagnostic Test: Nasal and Bronchial Sampling

INTERVENTIONS:
Diagnostic Test: Nasal and Bronchial Sampling — Nasal Absorption sampling, Bronchial sampling, Nasal Pharageal Aspirates, Blood sampling.

SUMMARY:
This study will compare the novel methods of NS and BS with the standard technique of nasophayngeal aspiration (NPA) and routine ETT suction. We shall assess the samples for diagnosis of RSV, viral load and immune responses in the airways of babies with RSV infection. We shall also assess the genetics of babies included in this study, to see if they may be vulnerable to RSV infection.

DETAILED DESCRIPTION:
In conjunction with a specialist medical device manufacturing company (Hunt Developments (Midhurst, West Sussex) we have produced novel nasosorption and bronchosorption kits that have CE marking. Both nasosorption and bronchosorption methods use synthetic absorptive matrix (SAM) strips: that look and feel like blotting paper, and will be placed onto the mucosal surface. These are comfortable to use and can be used at frequent intervals over extended periods of time. This non-invasive technique is ideal for infants and children, and it is possible to obtain neat mucosal lining fluid (MLF) even from normal healthy noses. The eluates contain cytokines and chemokines at high detectable levels on multiplex immunoassay.

We would like to use these SAMs to take MLF samples from the nasal and bronchial mucosal surfaces to see if these novel techniques can overcome the problems with current sampling methods. We plan to use these absorption techniques to measure RSV viral load. We also aim to look at the immune response in terms of the anti-viral interferon response (IFN-γ, IFN-λ, IFN-α2a, IP10, ITAC). In therapeutic studies in the future, it may be possible to document levels of drug (pharmacokinetics) in nasal MLF.

ELIGIBILITY:
Group 1 and Group 2

Inclusion Criteria

* Infants aged 2 weeks-24 months
* Presentation to the Emergency Department with any upper respiratory tract infection (URTI) in the RSV season (Oct-March).

OR • Documented RSV infection, admitted to the paediatric wards at St Mary's Hospital.

Exclusion Criteria

* Any local or systemic factor that would influence the safety of nasal sampling.
* Bilateral indwelling nasal catheters or local nasal pathology preventing access for nasal sampling.
* Bleeding disorders.
* The baby is taking part in another interventional study.
* The parents or guardians not able to sign the informed consent from due to limited English or comprehension despite the use of independent interpreter services.
* Limited life expectancy of the baby,

Group 3

Inclusion criteria

* Hospitalised Infants admitted to the PICU at St. Mary's Hospital, aged 2 weeks-24 months with documented RSV infection (by rapid test and/or PCR).
* Infants of weight >2kg.
* On a conventional ventilator with an Endotracheal Tube (ETT) of >3.0mmm diameter

Exclusion criteria

* Any local or systemic factor that would influence the safety of nasal sampling.
* Bilateral nasal catheters or local nasal pathology preventing access for nasal sampling.
* The baby is taking part in another interventional study.
* Prematurity - corrected gestational age <36 weeks, weight <2kg
* Significant hypoxia or instability precluding ventilator disconnection
* ETT < 3mm internal diameter
* Transcutaneous oxygen saturation of <95% on 60% oxygen
* Risk of bleeding
* Pneumothorax
* Infants receiving oral corticosteroid therapy at any time in past month
* Parents or guardians not able to sign informed consent from due to limited English or understanding despite the use of independent interpreter services.
* Limited life expectancy or a decision to limit management,

Control Group 1 Inclusion criteria

• Babies, aged 2 weeks-24 months, attending routine outpatient appointments or undergoing elective surgical procedures.

Exclusion criteria

* Any respiratory symptoms
* All other exclusion are the same as Groups 1 and 2

Control Group 2

Inclusion criteria

* Infants aged 2 weeks-24 months.
* Infants ventilated on the PICU for any condition
* Confirmed RSV negative by PCR of respiratory tract samples

Exclusion Criteria

* All exclusions are the same as Group 3
* In addition - any concern about raised intracranial pressure

Ages: 2 Weeks to 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 152 (Actual)
Dates: Start 2015-10-02 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Imperial College NHS Healthcare Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Participants consented that blood or nasal samples taken during this study can be used in the future for any ethically-approved studies.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Emergency Department | Paediatric Wards | Paediatric Intensive Care | Health Controls | Controls in Paediatric Intensive Care
Started | 32 | 51 | 49 | 20 | 0
Completed | 32 | 51 | 49 | 20 | 0
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Controls in paediatric intensive care were sought but non recruited
Groups:
- Total: Total of all reporting groups
Arm/Group | Emergency Department | Paediatric Wards | Paediatric Intensive Care | Health Controls | Controls in Paediatric Intensive Care | Total
Number analyzed (Participants) | 32 | 51 | 49 | 20 | 0 | 152
Age, Continuous [Mean (Full Range); unit: days] | 212 [27 to 630] | 186 [23 to 571] | 168 [14 to 630] | 168 [33 to 313] |  | 176 [14 to 630]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 22 | 15 | 7 | 0 | 53
  Male | 23 | 29 | 34 | 13 | 0 | 99
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 |  | 0
  Asian | 4 | 12 | 5 | 2 |  | 23
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 |  | 0
  Black or African American | 7 | 6 | 5 | 2 |  | 20
  White | 15 | 21 | 33 | 10 |  | 79
  More than one race | 6 | 12 | 6 | 6 |  | 30
  Unknown or Not Reported | 0 | 0 | 0 | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 32 | 51 | 49 | 20 |  | 152

OUTCOME MEASURES:

1. Primary Outcome: The Number of Sampling Visits on Which Participants Are Willing to Undergo Nasosorption and/or NPA Sampling
Description: To determine the difference in tolerability of nasosorption compared to NPA by assessment of acceptance by infants and families. Samples were collected from participants up to twice daily throughout study involvement, as such each participant could have >1 sampling visits.
Time Frame: Throughout symptomatic respiratory infection, up to 1 month
Population: Parents asked at each sampling timepoint on willingness to continue with respiratory sampling, as either: 1) both nasosorption and NPA, 2) just nasosorption, 3) just NPA, 4) discontinue sampling. This analysis includes all non-sedated hospitalised participants as sedation would influence the tolerability of sampling as perceived by parents/carers.
Measure: Number; unit: Sampling visits
Units Other Than Participants: Number of individual sampling visits
Groups:
- Wards: None sedated participants recruited from general paediatric wards
- Emergency Department: Non-ventilated participants recruited from the emergency department
Arm/Group | Wards | Emergency Department
Number analyzed (Participants) | 51 | 32
Number analyzed (Number of individual sampling visits) | 169 | 64
Sampling visits
  Nasosorption and NPA samples | 124 | 60
  NPA only | 0 | 0
  Discontinue sampling (while remaining in hospital) | 0 | 0
  Nasosorption only | 45 | 4

2. Primary Outcome: Accuracy of Nasosorption for Viral Load Measurement
Description: To determine the difference in accuracy of nasosorption compared to NPA by assessment of level of viral load (measured by qPCR).
Time Frame: Throughout symptomatic respiratory infection, up to 1 month
Population: Spearman R score correlation between RSV viral load as measured by nasosorption and NPA. This analysis includes all RSV+ infants independent of recruitment group as no differences in correlation between sample type were anticipated between recruitment group.
Measure: Number; unit: Spearman R score
Units Other Than Participants: Number matched RSV+ nasosorption and NPA
Groups:
- All Participants: Correlation between measurements of viral load and cytokines between nasosorption and NPA samples
Arm/Group | All Participants
Number analyzed (Participants) | 152
Number analyzed (Number matched RSV+ nasosorption and NPA) | 44
Spearman R score | 0.692

3. Secondary Outcome: Immune Response
Description: Establishing the use of nasal and bronchial sampling to measure the host immune response to RSV. We will determine cytokine and inflammatory mediator concentrations by immunoassay of eluted fluid from nasosorption and compare with NPA.
Time Frame: Throughout symptomatic respiratory infection, up to 1 month
Population: Spearman R score correlation of Interferon-gamma levels in matched nasosorption and NPA samples from any participant. This analysis includes all RSV+ infants independent of recruitment group as no differences in correlation between sample type were anticipated between recruitment group.
Measure: Number; unit: Spearman R score
Units Other Than Participants: Number matched nasosorption and NPA
Groups:
- All Participants: Correlation between measurements of cytokines (exemplified by Interferon-gamma) between nasosorption and NPA samples
Arm/Group | All Participants
Number analyzed (Participants) | 152
Number analyzed (Number matched nasosorption and NPA) | 124
Spearman R score | 0.0001

4. Primary Outcome: Accuracy of Bronchosorption for Viral Load Measurement, Compared to Tracheal Aspirate
Description: To determine the difference in accuracy of bronchosorption (BSAM) compared to tracheal aspirate (TA) by assessment of level of viral load (measured by qPCR).
Time Frame: Throughout symptomatic respiratory infection, up to 1 month
Population: Spearman R score correlation between RSV viral load as measured by bronchosorption and tracheal aspiration. This analysis includes all RSV+ infants independent of recruitment group as no differences in correlation between sample type were anticipated between recruitment group.
Measure: Number; unit: Spearman R score
Units Other Than Participants: Number matched RSV+ BSAM and TA
Arm/Group | All Participants
Number analyzed (Participants) | 24
Number analyzed (Number matched RSV+ BSAM and TA) | 20
Spearman R score | 0.45

ADVERSE EVENTS:
Time Frame: Throughout participant hospitalisation, to a maximum of 6 months after the end of sampling
Description: As per clinicaltrials.gov definitions
Arm/Group | Emergency Department | Paediatric Wards | Paediatric Intensive Care | Health Controls | Controls in Paediatric Intensive Care
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/51 | 0/49 | 0/20 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/51 | 0/49 | 0/20 | 0/0
Other Adverse Events (participants affected / at risk) | 0/32 | 0/51 | 0/49 | 0/20 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-17): https://cdn.clinicaltrials.gov/large-docs/17/NCT03062917/Prot_SAP_000.pdf